CLINICAL TRIAL: NCT05719623
Title: Effects of Cuevas Medek Exercises on Balance and Postural Control in Children With Spastic Cerebral Palsy
Brief Title: Cuevas Medek Exercises on Balance and Postural Control in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0734
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Spastic Cerebral Palsy
Keywords: Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Postural Balance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CUEVAS MEDEK EXERCISES (Experimental): Experimental group will get conventional treatment along with Cuevas Medak Exercises
  Interventions: Other: CUEVAS MEDEK EXERCISES
- BALANCE AND POSTURAL (Other): Controlled will get conventional treatment
  Interventions: Other: BALANCE AND POSTURAL

INTERVENTIONS:
Other: CUEVAS MEDEK EXERCISES — stretchings/strengthening
  Other Names: Conventional Physical therapy
  Arms: CUEVAS MEDEK EXERCISES
Other: BALANCE AND POSTURAL — BALANCE AND POSTURAL
  Arms: BALANCE AND POSTURAL

SUMMARY:
Cerebral palsy (CP) is a disorder characterized by abnormal tone, posture and movement and clinically classified based on the predominant motor syndrome-spastic hemiplegia, spastic diplegia, spastic quadriplegia, and extra-pyramidal or dyskinetic. Clinical prediction models and neuroimaging have been used to diagnose CP before the age of 2 years, but further research is necessary. Cuevas Medek Exercises (CME) is a pediatric physiotherapy approach for children with developmental motor delay impacting the central nervous system. According to Ramon Cuevas, who developed the therapy, CME are mainly based on the principle of provoking novel automatic motor reactions using exercises against gravity with progressive distal holding. This study will find the effects of Cuevas Medak Exercises on Balance and Postural control in children with spastic cerebral palsy.

This Randomized Controlled Trial will recruit the participants through random sampling. Participants will be randomly divided into 2 groups. Two groups of children aged between 2 and 5 years, suffering from cerebral palsy in spastic form, one for control and one for experiment. Controlled will get conventional treatment while study group will get conventional treatment with Cuevas Medak Exercises. Treatment duration is of 12 weeks. Progress will monitored every month. The frequency of recovery sessions will 3 sessions/week, and the duration of a session will 45 minutes. Patient evaluation will be made at the beginning and the end of the treatment through pediatric balance scale and static balance test. Data will be analyzed through SPSS 25.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a disorder characterized by abnormal tone, posture and movement and clinically classified based on the predominant motor syndrome-spastic hemiplegia, spastic diplegia, spastic quadriplegia, and extra-pyramidal or dyskinetic (1). Children born preterm account for one-third to one-half of CP diagnoses in HICs, although this proportion is much lower in low-income countries (LICs), where mortality of very preterm babies remains high . Clinical prediction models and neuroimaging have been used to diagnose CP before the age of 2 years, but further research is necessary (.

The CPs share a common clinical sign of non-progressive dysfunction of posture and movement control but not a common diagnosis. Although there are many CP types, many causes, and now many associated pathogenic genetic variants, it is probably not advisable to change the clinical diagnosis of CP made by specialist pediatricians in cases that fulfill the clinical definition.

In order to prevent greater developmental motor delay, a physiotherapy intervention focusing on optimizing neuroplasticity must be done, stimulating the child to achieve the developmental motor milestones . Cuevas Medek Exercises (CME) is a pediatric physiotherapy approach for children with developmental motor delay impacting the central nervous system. According to Ramon Cuevas, who developed the therapy, CME are mainly based on the principle of provoking novel automatic motor reactions using exercises against gravity with progressive distal holding CME therapy is a physiotherapy approach to treat children with developmental motor delay by impacting CNS. Postural control and balance training are essentials for the children to be mobile. The aim of the study is to find the effects of Cuevas Medek Exercises on balance and postural control on children with spastic Cerebral Palsy so that the children with motor development disorders of neurological cause like cerebral palsy can develop automatic motor reactions which they would not be able to develop on their own, because of neurological injuries and help them to improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Children with medical diagnosis of Spastic Cerebral Palsy
* Age ranging from 2 to 5 years.
* Children who will able to stand and walk

Exclusion Criteria:

* Children with planned surgical or medical surgeries during study period
* Children with impaired cognition
* Children with hearing impairment and visual impairment

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
pediatric balance scale | 12 weeks
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points

SECONDARY OUTCOMES:
static balance test. | 12 weeks
  The Four Stage Balance Test is a validated measure recommended to screen individuals for fall risk. It is based on the persons ability to hold four progressively more challenging positions[1](evaluates static balance).

CONTACTS AND LOCATIONS:
Overall Officials: Sara khan, MS, Principal Investigator — Riphah International University
Locations (1):
- Helping Hands Organization (HHRD) Bahawalpur., Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No